CLINICAL TRIAL: NCT00036998
Title: A Randomized Pivotal Clinical Trial In Breast Cancer Patients Of Pre-Operative Focal Microwave Thermotherapy Treatment For Early-Stage Breast Disease In Intact Breast
Brief Title: Microwave Thermotherapy in Treating Women With Stage I or Stage II Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imunon (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069347; CELSION-10200202; OU-09532
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2004-07

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

INTERVENTIONS:
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Procedure: thermal ablation therapy

SUMMARY:
RATIONALE: Microwave thermotherapy kills tumor cells by heating them to several degrees above body temperature.

PURPOSE: Randomized phase II trial to compare the effectiveness of microwave thermotherapy before surgery to that of surgery alone in treating women who have stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the safety and efficacy of preoperative focused microwave thermotherapy followed by surgery vs surgery alone in women with early-stage primary breast cancer.
* Compare the reduction of tumor cells at surgical margins and second incision rates in women treated with these regimens.
* Compare the percentage of pathological cell death in women treated with these regimens.
* Compare the amount of surgically removed breast and tumor tissue in women treated with these regimens.
* Compare the measurement of the extent tumor margins of the surgically removed breast and tumor tissue in women treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to tumor classification (T1 vs T2) and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I:Patients undergo ultrasound-guided placement of a microwave sensor and a temperature probe (before or after compression of the breast) and external placement of 2 large opposing microwave emitters and up to 7 skin temperature sensors on the compressed breast. Patients then receive focused microwave thermotherapy that slowly heats the primary breast tumor and deep proximal breast tissue. In the absence of undue heating of the skin, a tumor temperature of 48-52° C is targeted and maintained for an equivalent thermal dose of 140-180 minutes.

Within 60 days of thermotherapy, patients undergo lumpectomy.

* Arm II: Patients undergo lumpectomy only. Patients are followed at 30 and 90 days after surgery, and then at the discretion of the physician.

PROJECTED ACCRUAL: A total of 200-222 patients (100-111 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary breast cancer by core needle biopsy

  * T1a, b, c, or T2
  * Diagnosis not made with a lumpectomy or incisional biopsy
* Candidate for breast conservation surgery (lumpectomy/radiotherapy)
* Tumor measurable by breast ultrasound
* No metastatic disease, including skin metastases
* No bilateral breast cancer
* No high-probability of extensive intraductal disease in situ
* No clinical fixation to the pectoralis major muscle or skin
* No involvement of the nipple
* No inflammatory breast cancer
* No multicentric disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 6 months

Hematopoietic:

* Platelet count at least 100,000/mm^3 (no thrombocytopenia)
* No bleeding disorders

Hepatic:

* PT, INR, and PTT less than 1.5 times normal
* Bilirubin no greater than 2.0 mg/dL
* Transaminases no greater than 2 times normal
* No coagulopathy
* No liver disease

Renal:

* BUN less than 30 mg/dL
* Creatinine less than 1.9 mg/dL
* No renal insufficiency

Cardiovascular:

* No pacemakers or defibrillators
* No clinically significant heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of effective contraception, including 1 barrier method
* Able to tolerate prone position and breast compression
* No breast implants
* No prior collagen vascular disease
* No other factor or condition (other than tumor size) that would preclude lumpectomy
* No mental condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Other:

* No prior participation in this study
* More than 30 days since prior participation in another clinical study
* No concurrent anticoagulants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-08

CONTACTS AND LOCATIONS:
Overall Officials: William E. Gannon, MD, Study Chair — Imunon
Locations (8):
- United States (7):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Comprehensive Breast Center of Coral Springs, Coral Springs, Florida
  - Oklahoma University Medical Center at University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mroz-Baier Breast Care Center, Memphis, Tennessee
  - Breast Care Specialists, P.C., Norfolk, Virginia
  - Tacoma, Washington
- Royal Bolton Hospital, Bolton, Lancashire, England, United Kingdom